CLINICAL TRIAL: NCT07205016
Title: FreeFrail Project: Effectiveness of a Multicomponent Intervention Including Dual-task Exercise to Increase Functionality and Cognitive Performance in Frail and Pre-frail Individuals Over 65 Years Aged in Primary Care Compared to Usual Care: Protocol for a Randomized Controlled Trial
Brief Title: FreeFrail Project: A Multicomponent Intervention for the Management of Frailty in Primary Care: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Oriol Martínez Navarro, Doctor, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FreeFrail Project
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Frail Elderly; Dual Task Exercises in Elderly People; Exercise Training; Frailty
Keywords: primary care Health [MeSH]; multicomponent intervention; exercise therapy [MeSH]; cognitive-motor dual-task; frail elderly [MeSH]; frailty [MeSH]
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, parallel-group controlled trial will be conducted in primary care centers in Lleida
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The intervention group will conduct the same multicomponent intervention than the control group, but adding the dual cognitive task while performing the therapeutic physical activity, which may include counting numbers backwards, in 2s, mentioning names of animals, food, countries and others. The objective of this additional condition is to stimulate cognitive and functional capacity simultaneously, increasing the complexity of the activity and the transfer to daily life activities
  Interventions: Behavioral: Dual task exercise
- Control (Active Comparator): A multicomponent program designed to address frailty in community-dwelling older adults. It integrates three evidence-based domains: therapeutic physical activity, cognitive psychological intervention, and nutritional support.
  The three components are delivered in a coordinated manner by a multidisciplinary team at ICS. Intervention fidelity is ensured through standardized protocols, training of professionals, and monitoring of adherence.
  The therapeutic physical activity program will be structured across three progressive levels-beginner, intermediate, and advanced-to accommodate varying functional capacities. Strength training will advance through incremental increases in repetitions and resistance, while balance exercises will become more challenging by reducing external support. The material for the session will be in the same room where the group is held and will include the use of weights or dumbbells, elastic bands, balls, and pikes
  Interventions: Behavioral: Otago exercise

INTERVENTIONS:
Behavioral: Dual task exercise — The intervention group will conduct the same multicomponent intervention than the control group, but adding the dual cognitive task while performing the therapeutic physical activity, which may include counting numbers backwards, in 2s, mentioning names of animals, food, countries and others. The objective of this additional condition is to stimulate cognitive and functional capacity simultaneously, increasing the complexity of the activity and the transfer to daily life activities.
  Arms: Experimental
Behavioral: Otago exercise — The proposed intervention is a multicomponent program designed to address frailty in community-dwelling older adults. It integrates three evidence-based domains: therapeutic physical activity, cognitive psychological intervention, and nutritional support.
  Arms: Control

SUMMARY:
The primary aim is to assess the effectiveness of a multicomponent intervention including dual-task exercise in improving functionality and cognitive performance and in reducing frailty among community-dwelling adults aged ≥65 years compared to usual care. Secondary objectives include evaluating its impact on pain, anxiety or depression, sleep quality, quality of life, physical activity, handgrip strength, and polypharmacy.

A double-blind, randomized, parallel-group controlled trial will be conducted in primary care centers in Lleida. Frail older adults (≥65 years) will be recruited and randomly allocated to either the intervention group, receiving a structured cognitive-motor dual-task based multicomponent program, or the control group, receiving usual care. Outcomes will be assessed using validated tools at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Frailty according to Fragil-VIG index (>0,20)
* Barthel index > 60
* Able to perform physical exercise
* Able to understand and communicate in Catalan or Spanish

Exclusion Criteria:

* Decompensated / Unstable cardiovascular disease or recent diagnosed
* Upper or lower injury with functional impairment
* Institutionalized patient.
* Terminal or tumoral processes
* People who participated in another clinical trial or exercise programme during last year
* Diagnosis of severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Physical performance and functional status | From enrollment to the end of treatment at 12 weeks
  The Short Physical Performance Battery (SPPB) is an ordinal quantitative scale ranging from 0 to 12. This validated tool assesses three functional domains: lower-limb muscle strength, by timing the repeated chair-stand test; gait speed, through the 4-meter walking test; and static balance, evaluated with three progressively difficult positions (feet together, semi-tandem, tandem). A composite score is calculated, with lower values reflecting poorer performance. A score of 9 or less has been widely adopted as a cut-off point for identifying frailty and pre-frailty in older adults, making this instrument particularly suitable for evaluating the effectiveness of interventions on physical function
Cognitive function | From enrollment to the end of treatment at 12 weeks
  The Mini-Mental State Examination (MMSE) is a continuous quantitative widely used 30-point screening tool validated for older adults to assess global cognitive function. It evaluates orientation, memory, attention, language, and praxis, providing a standardized quantitative measure of cognitive status. Although limited in sensitivity for mild or executive deficits, the MMSE remains a practical first-line assessment in frailty research and clinical protocols, and its integration alongside multidimensional frailty measures allows for a more comprehensive characterization of cognitive vulnerability in aging. A culturally adapted and validated version is available in Spanish, enabling its use in Hispanic populations.
Frailty status | From enrollment to the end of treatment at 12 weeks
  The Frailty-VIG is an ordinal quantitative measure specifically validated for older adults in the community. This multidimensional tool comprises 22 dichotomous items spanning activities of daily living, nutrition, cognition, emotional health, social context, geriatric syndromes, and chronic diseases. By incorporating multimorbidity and psychosocial domains alongside physical aspects, the Frailty-VIG provides a comprehensive assessment of frailty, overcoming the limitations of purely physical indices

SECONDARY OUTCOMES:
Quality of life / Anxiety and Depression / Pain severity | From enrollment to the end of treatment at 12 weeks
  will be evaluated with the EuroQoL-5D-5L which generates ordinal categorical variables from five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-point Likert scale, where higher scores denote lower quality of life. This standardized and validated instrument has been extensively applied in Spanish populations and is particularly appropriate to capture the multidimensional impact of frailty on health-related quality of life
Sleep performance | From enrollment to the end of treatment at 12 weeks
  will be assessed using the Spanish validated version of the Pittsburgh Sleep Quality Index (PSQI). This self-administered questionnaire yields a global score between 0 and 21, with higher scores reflecting worse sleep quality. It evaluates seven components-subjective quality, latency, duration, habitual efficiency, disturbances, medication use, and daytime dysfunction. A score above 5 is commonly considered indicative of clinically relevant sleep impairment. As poor sleep has been consistently associated with frailty and functional decline, the PSQI offers a sensitive and appropriate measure for this study
Physical activity | From enrollment to the end of treatment at 12 weeks
  will be assessed through the International Physical Activity Questionnaire (IPAQ), which produces continuous quantitative data expressed in metabolic equivalent task minutes per week (MET-min/week). It includes seven open questions regarding activity over the previous seven days, covering walking, moderate and vigorous activities, and sedentary behaviour. The calculation of MET-min/week allows standardized estimation of global activity levels. This questionnaire is validated and widely used in community-dwelling adults, making it an appropriate measure for capturing the impact of the intervention on activity levels
Handgrip strength | From enrollment to the end of treatment at 12 weeks
  will be measured with a handheld dynamometer. Results are expressed as continuous quantitative variables in kilograms. Following standardized protocols, participants will be seated with the elbow flexed at 90° and the wrist positioned between neutral and 30° dorsiflexion. They will be instructed to squeeze the dynamometer maximally for 3-5 seconds. Three trials will be performed alternately in each hand, with one-minute rest intervals, and the best value will be recorded. Handgrip strength is a simple, reliable, and validated marker of sarcopenia and frailty risk, strongly correlated with morbidity and mortality in older adults
Inflammatory and mitochondrial function biomarkers | From enrollment to the end of treatment at 12 weeks
  are strongly supported by the literature in frail population, as these biological factors are fundamentally implicated in the pathways leading to frailty, sarcopenia, and functional impairment. Chronic low-grade inflammation ("inflammaging"), a hallmark of aging, is characterized by increased levels of circulating pro-inflammatory cytokines such as interleukin 6 and 8(IL-6, IL-8), interleukin 1β (IL-1β), tumor necrosis factor-α (TNF-α), and C-reactive protein (CRP). These biomarkers consistently correlate with chronic low-grade inflammation ("inflammaging") and mitochondrial dysfunction (3) they have also been consistently associated with sarcopenia, frailty, and functional decline (4,5) . The blood samples will be analysed at Biomedical Research Institute of Lleida (IRB Lleida), generating continuous quantitative data.

IPD SHARING:
Plan to Share IPD: Undecided